CLINICAL TRIAL: NCT05075512
Title: A Prospective Study on Efficacy and Safety of Anlotinib Combined With Fulvestrant in Patients With HR-positive and HER2-negative, Secondary Endocrine-resistant, Locally Advanced or Metastatic Breast Cancer
Brief Title: The Efficacy and Safety of Anlotinib Combined With Fulvestrant in Patients With Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021SQGH00743
Record Dates: First submitted 2021-08-09; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — anlotinib; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): anlotinib combined with fulvestrant
  Interventions: Drug: anlotinib, fulvestrant

INTERVENTIONS:
Drug: anlotinib, fulvestrant — anlotinib: 12 mg once daily on days 1-14, repeated every 21 days; fulvestrant: 500 mg on days 1 and 15 of cycle one, and then on day one of each subsequent 28 days cycle
  Other Names: AL3818

SUMMARY:
The management of HR-positive, HER2-negative metastatic breast cancer includes endocrine monotherapy or combination regimens, both with benefit diminishing as resistance develops. Nowadays, various studies have demonstrated that estrogen interacts with many angiogenic pathways and is an important mechanism for resistance leading to the question of whether combination with antiangiogenesis and antiestrogen therapies could be an appropriate therapeutic modality. Anlotinib is a novel multi-target tyrosine kinase inhibitor that effectively inhibit VEGFR, FGFR, PDGFR, c-KIT, c-MET and RET. Previous studies have proven the efficacy of both anlotinib monotherapy and combination regimens in advanced breast cancer. This phase II study aims to preliminarily evaluate the efficacy and safety of anlotinib combined with endocrine therapy.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label, phase II clinical trial. The secondary endocrine-resistant is defined as disease relapse within 12 months after at least 24 months endocrine adjuvant therapy, or disease progress after at least 6 months endocrine salvage therapy. Eligible patients were treated with oral anlotinib plus intramuscular fulvestrant till disease progression or intolerant toxicity. In the part of statistical analysis, 40 patients are required to have a 80% power to detect significant improvement in median progression-free survival from 5.8 (fulvestrant alone) to 10 (fulvestrant combined with anlotinib) months, if tested at a two-sided significance level of α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older female；
* ECOG score 0-1;
* Life expectancy is not less than 12 weeks;
* Histology confirmed HR-positive and HER2-negative locally advanced or metastatic breast cancer;
* Premenopausal women have taken effective ovarian function suppression methods, such as drug suppression or ovariectomy;
* At least one objectively measurable breast cancer lesions according to RECIST 1.1 ;
* No more than one systemic chemotherapy for metastatic disease;
* Disease relapse within 12 months after at least 24 months endocrine adjuvant therapy, or disease progress after at least 6 months endocrine salvage therapy;
* Normal function of main organs and bone marrow: Hemoglobin≥90g/L; Neutrophil count (ANC)≥1.5×109/L; Platelet count (PLT)≥80×109/L; Total bilirubin≤1.5×ULN (upper limit of normal); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (≤5×ULN if has liver metastasis); Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60mL/min (Cockcroft-Gault formula);
* Sign the informed consent;

Exclusion Criteria:

* Have received prior fulvestrant or anti-angiogenic drug treatment, or known to be allergic to any excipients in the study;
* Visceral crisis;
* Uncontrolled or high-burden CNS metastases;
* Unable to swallow;
* Abnormal coagulation function;
* Tumor has invaded important blood vessels and may cause fatal bleeding;
* Pleural effusion or pericardial effusion that requiring repeated drainage;
* Hypertension that cannot be well controlled by a single antihypertensive drug;
* Unstable angina, myocardial infarction within 6 months, serious arrhythmias;
* The history of immunodeficiency, including HIV or other obtained or congenital immunodeficiency diseases, or a history of organ transplantation;
* Poorly controlled diabetes;
* Abnormal urine protein, and the 24-hour quantification suggests urine protein ≥1.0g;
* Bleeding constitution or medical history
* Unhealed wounds, ulcers or fractures;
* Have arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
* In other clinical trials of anti-tumor drugs simultaneously;
* Other concomitant disease or disability that endangers safety according to the judgment of investigator;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From randomisation to progression or death, assessed up to 60 months
  Time from randomisation to tumour progression (in any way) or death (from any cause)

SECONDARY OUTCOMES:
Overall Response Rate | From randomisation to the first occurrence of the confirmed complete response or partial response, assessed up to 24 months
  Confirmed complete response or partial response according to RECIST 1.1
Clinical Benefit Rate | From randomisation to the first occurrence of the confirmed complete response or partial response or stable disease, assessed up to 24 months
  Confirmed complete response or partial response or stable disease of 24 weeks' duration or longer
Overall Survival | From randomisation to death, assessed up to 96 months
  Time from randomisation to death (from any cause)
Adverse events | From randomisation to 30 days after the last dose administrated
  Adverse events occurred from randomisation to 30 days after the last dose administrated

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
the data will be shared from the trial begin and for 10 years
Supporting Information: Study Protocol, SAP, CSR
Time Frame: from the trial begin and for 10 years
Access Criteria: every one